CLINICAL TRIAL: NCT06772857
Title: Aerobic Versus Resistance Exercises on Insulin Sensitivity in Obese Patients
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: National Police Hospital (Other Government)
Responsible Party: Principal Investigator, El-Sayed Essam, Lecturer at Department of Physical Therapy for Cardiovascular/Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004665
Record Dates: First submitted 2024-12-29; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Insulin Sensitivity/Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: The purpose of study is to compare the effect of different exercise modes on insulin resistance and body composition in obese patients
Who Masked: Care Provider
Masking Description: Study group A (20 patients):will receive aerobic exercise training in addition to medical and diet regimen. This mode of exercise training will be applied 3 times/week for six weeks.
  Study group B (20 patients): will receive resistance exercise training in addition to medical and diet regimen. This mode of exercise training will be applied 3 times/week for six weeks.
  Control group C (20 patients): will receive medical and diet regimen only for six weeks. The patients will be instructed not to change their physical activity during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A: Aerobic Exercise + Medical and Diet Regimen (Experimental): Study group A (20 patients) will receive aerobic exercise training in addition to a medical and diet regimen. Aerobic exercise training will be applied 3 times per week for 6 weeks. This exercise will include activities such as walking, cycling, or swimming to improve cardiovascular fitness and insulin sensitivity.
  Interventions: Drug: Metformin
- Group B: Resistance Exercise + Medical and Diet Regimen (Experimental): Study group B (20 patients) will receive resistance exercise training along with a medical and diet regimen. Resistance exercise training will be applied 3 times per week for 6 weeks, focusing on strength-building exercises to improve muscle mass and insulin sensitivity.
  Interventions: Drug: Metformin
- Group C: Medical and Diet Regimen Only (Active Comparator): Control group C (20 patients) will receive only a medical and diet regimen for 6 weeks. Patients in this group will be instructed not to change their physical activity during the study period.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin is a drug used to manage blood glucose levels. It improves insulin sensitivity and reduces glucose production in the liver. This regimen will be provided to all study groups (A, B, and C) in combination with the respective interventions described for each group. Participants are instructed not to change their physical activity during the study.
  Other Names: Glucophage; Glucophage XR; Riomet

SUMMARY:
The purpose of study is to compare the effect of different exercise modes on insulin resistance and body composition in obese patients.

DETAILED DESCRIPTION:
The global epidemic of obesity becomes a major healthy, social, and economical burden.Indeed, it has been well established that obesity directly increases cardio metabolic risk by altering the insulin sensibility. Moreover, obesity causes additional health problems as it is closely associated with the development and progression of coronary heart disease.

According to the World Health Organization (WHO), Egypt ranks 18th with the highest prevalence of obesity worldwide.( Global Obesity Levels,2020) Deaths attributable to non-communicable diseases represent about 71% of the total mortality burden .(World Health Organization,2021) Lack of exercise and sedentary behaviour (prolonged sitting) are major risk factors for insulin resistance The prevalence of obesity has increased in adults in Egypt to reach about 40% according to 100million health survey (2019) compared to the 36% estimate of 2017 STEPwise survey .

This review presents established knowledge on the effects of physical activity (PA) on whole-body insulin sensitivity (SI) and body composition .

1. Sixty obese prediabetic patients from both sexes with ages ranging from 30 to 40 years old.
2. Their body mass index will be ranged from 30 to 34.9 kg/m2.
3. They have insulin resistance assessed by the homeostasis model assessment for insulin resistance (HOMAIR) Levels above 1.9
4. Their blood glucose level will be ranged from 100 to 125 mg/dL (5.6-6.9 mmol/l)
5. They will receive the same medical and diet regimen in addition to instructions not to change their physical activity during the study.

Study group A (20 patients):will receive aerobic exercise training in addition to medical and diet regimen. This mode of exercise training will be applied 3 times/week for six weeks.

Study group B (20 patients): will receive resistance exercise training in addition to medical and diet regimen. This mode of exercise training will be applied 3 times/week for six weeks.

Control group C (20 patients): will receive medical and diet regimen only for six weeks. The patients will be instructed not to change their physical activity during the study.

ELIGIBILITY:
Inclusion Criteria:

* Sixty obese prediabetic patients from both sexes with ages ranging from 30 to 40 years old.
* Body mass index (BMI) ranging from 30 to 34.9 kg/m².
* Insulin resistance as assessed by the homeostasis model assessment for insulin resistance (HOMA-IR) levels above 1.9.
* Blood glucose levels ranging from 100 to 125 mg/dL (5.6-6.9 mmol/L).
* Patients will receive the same medical and diet regimen, with instructions not to change their physical activity during the study.
* HbA1c levels between 6.0% and 6.5%, indicating high risk for diabetes and possible consideration for prevention interventions.

Exclusion Criteria:

* Uncontrolled diabetes.
* Uncontrolled hypertension.
* Cardiovascular disease.
* Respiratory disease.
* Hepatic disease.
* Severe life-limiting illness (e.g., cancer).
* Use of weight loss medications.
* Orthopedic or neurological disorders that limit exercise participation.
* Endocrine disorders.
* Kidney disease.

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Insulin Resistance Between Different Exercise Modes in Obese Patients | 3months
  The change in insulin resistance will be assessed using the HOMA-IR index in obese patients after different exercise interventions (aerobic vs resistance) compared to baseline. The HOMA-IR index will be calculated based on fasting blood glucose and fasting insulin levels, which are widely accepted measures of insulin resistance.

CONTACTS AND LOCATIONS:
Overall Officials: El-sayed Felaya, Principal Investigator — Respiratory Disorder and Geriatrics Faculty of Physical Therapy Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No